CLINICAL TRIAL: NCT06376942
Title: A Randomized, Double-blind, Placebo-controlled Trial to Compare the Effectiveness of Nebulized Anticholinergics for Cough Suppression During Flexible Bronchoscopy
Brief Title: A RCT to Compare the Effectiveness of Nebulized Anticholinergics for Cough Suppression During Flexible Bronchoscopy
Acronym: NAFCOF
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ritesh Agarwal, Professor of Pulmonary Medicine, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Int/IEC/2024/SPL-5
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Subjects Undergoing Flexible Bronchoscopy
MeSH Terms: interventions — Glycopyrrolate; Ipratropium; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Glycopyrronium (Experimental): Nebulized glycopyrronium 50 mcg (2 ml) administered via a jet nebulizer over 10 minutes
  Interventions: Drug: Glycopyrronium
- Ipratropium (Active Comparator): Nebulized ipratropium bromide 500 mcg (2 ml) administered via a jet nebulizer over 10 minutes
  Interventions: Drug: Ipratropium
- Saline (Placebo Comparator): Nebulized saline 0.9% (2 ml) administered via a jet nebulizer over 10 minutes
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Glycopyrronium — Nebulized glycopyrronium 50 mcg
  Arms: Glycopyrronium
Drug: Ipratropium — Nebulized iptratropium 500 mcg
  Arms: Ipratropium
Other: Saline — 0.9% saline 2 ml
  Arms: Saline

SUMMARY:
No study has examined the role of inhaled glycopyrrolate on mucus secretion. We hypothesize that nebulized glycopyrrolate will improve bronchoscopy procedure by effectively suppressing airway mucus secretion, thereby decreasing cough, and thus improving patient comfort during bronchoscopy. In this study, we aim to compare the efficacy of nebulized glycopyrrolate versus nebulized ipratropium in suppression of cough during flexible bronchoscopy.

DETAILED DESCRIPTION:
Bronchoscopy is a minimally invasive endoscopic technique for direct visualization of airways, with diagnostic and therapeutic intent. In 1897, Killian laid the foundation of bronchoscopy by extracting an animal bone from the right main bronchus of a farmer using rigid esophagoscope. In 1966, Shigeto Ikeda developed a prototype of flexible bronchoscope. Since its inception, flexible bronchoscope has undergone advancements in design and technology. The technological advancements in the recent decades have improved diagnostic yield and safety, with low morbidity and mortality. Unfortunately, the occurrence of cough during flexible bronchoscopy makes the procedure difficult and increases procedure time with patient discomfort.

Owing to the lack of clinical benefits and possible hemodynamic changes, the British Thoracic Society and Joint Indian Chest Society recommend not to use anticholinergic premedication via the parenteral route for preventing cough before bronchoscopy.

bronchoscopy. A few studies have evaluated inhaled anticholinergic premedication. Inoue et al. (in 1994) studied the effects of inhaled ipratropium bromide on bronchoconstriction in 29 subjects underwent for diagnostic bronchoscopy. They concluded that ipratropium protects against the deleterious effects resulting from topical lidocaine anesthesia during bronchoscopy. Wang et al. evaluated the efficacy of ipratropium bromide in 250 patients in a placebo-controlled trial. They reported that nebulized ipratropium bromide could reduce airway secretions and patient discomfort.

To our knowledge, no study has examined the role of inhaled glycopyrrolate on mucus secretion. We hypothesize that nebulized glycopyrrolate will improve bronchoscopy procedure by effectively suppressing airway mucus secretion, thereby decreasing cough, and thus improving patient comfort during bronchoscopy.

In this study, we aim to compare the efficacy of nebulized glycopyrrolate versus nebulized ipratropium in suppression of cough during flexible bronchoscopy.

ELIGIBILITY:
Inclusion Criteria: Consecutive patients with indication for flexible bronchoscopy will be enrolled in the study if they meet all the following criteria:

* age ≥18 years
* hemodynamically stable
* willing to provide a written informed consent

Exclusion Criteria: Patients with any of the following will be excluded:

* intubated or tracheostomized patients
* patients with airway stent in situ
* patients with a history of glaucoma
* baseline oxygen saturation <90%
* patients with hemodynamic instability (SBP <90 mm Hg)
* patients undergoing sedation for bronchoscopy
* failure to provide informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2024-04-24 (Estimated); Primary Completion 2025-04-25 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Cough count | Intra-procedure
  Objectively measured using condenser microphone and voice recording application though a smartphone

SECONDARY OUTCOMES:
Operator-estimated airway secretion | Intra-procedure
  Recorded as: almost none, needing saline to wash out, and excessive, making it difficult to visualize the airways and requires 5 ml aliquots of saline
Operator-rated secretions on a visual analogue scale (VAS) | Immedidate post-procedure
  100 mm VAS anchored as no secretion at one and maximal secretions at the other
Operator-rated cough intensity on a visual analogue scale (VAS) | Immedidate post-procedure
  100 mm VAS anchored as no cough at one and maximal cough at the other
Patient-rated comfort on a visual analogue scale (VAS) | Immedidate post-procedure
  100 mm VAS anchored as maximal comfort at one and maximal discomfort at the other
Adverse reactions | 1-hour post-procedure
  Arrhythmia, glaucoma, nausea, headache

CONTACTS AND LOCATIONS:
Locations (1):
- Bronchoscopy suite, PGIMER, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No